CLINICAL TRIAL: NCT03868072
Title: An Open-label, Randomized, Fasted, Single Dose, Crossover Study to Evaluate the Bioequivalence of Chong Kun Dang Pharmaceutical "Chong Kun Dang Tofacitinib Tablet" and Pfizer Korea Inc. "XELJANZ 5Mg Tablet" in Healthy Volunteers
Brief Title: Study to Evaluate the Bioequivalence of Pfizer Korea Inc. "XELJANZ 5Mg Tablet" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BE118111814 / BN1-18-118
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference/Test (Experimental): 1. Period 1: XELJANZ 5Mg Tablet 1T
  2. Period 2: Chong Kun Dang Tofacitinib Tablet 1T
  Interventions: Drug: XELJANZ 5Mg Tablet; Drug: Chong Kun Dang Tofacitinib Tablet
- Test/Reference (Experimental): 1. Period 1: Chong Kun Dang Tofacitinib Tablet 1T
  2. Period 2: XELJANZ 5Mg Tablet 1T
  Interventions: Drug: XELJANZ 5Mg Tablet; Drug: Chong Kun Dang Tofacitinib Tablet

INTERVENTIONS:
Drug: XELJANZ 5Mg Tablet — XELJANZ 5Mg Tablet 1T single oral administration under fasting
Drug: Chong Kun Dang Tofacitinib Tablet — Chong Kun Dang Tofacitinib Tablet 1T single oral administration under fasting

SUMMARY:
This study is an open-label, randomized, fasted, single dose, crossover study to evaluate the bioequivalence of Chong Kun Dang Pharmaceutical "Chong Kun Dang Tofacitinib Tablet" and Pfizer Korea Inc. "XELJANZ 5Mg Tablet" in healthy volunteers

DETAILED DESCRIPTION:
To healthy subjects of forty (40), following treatments are administered dosing in each period and wash-out period is a minimum of 1 week.

Reference drug: XELJANZ 5Mg Tablet / Test drug: Chong Kun Dang Tofacitinib Tablet Pharmacokinetic blood samples are collected up to 12hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject older than 19 years at the screening
2. Individuals who had 18 kg/m2 ≤ Body Mass Index(BMI) ≤ 30kg/m2

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination(if necessary, EEG, ECG, chest X-ray, endoscope or upper gastrointestinal radiography)
4. Individuals who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, ECG, chest X-ray etc.)
5. Women who are not pregnant at physical examination

Exclusion Criteria:

1. Individuals who had enrolled to barbiturate's drugs by induction and inhibition of drug-metabolizing enzymes of drugs, such as drugs or excessive drinking within the 1 month
2. Individuals who had taken any medication within 10 days prior to the first day of dosing
3. Individuals who were deemed to be inappropriate to participate in the study by the investigator
4. Individuals who had participated of other clinical study or bioequivalence study within the 3 months prior to the first day of dosing
5. Individuals who donated whole blood within the 2 months, or blood components within 2 weeks prior to the first dose of the investigational product(s)
6. Individuals who do not agree to the approved methods of double contraception and using spermicide for up to 7 days (only, 4 weeks for women who may be pregnant) after investigational product(s) administration (Double contraception: two or more of the use of condoms, intrauterine contraception, diaphragm, cervical cap, or a sexual partner who had been medically diagnosed infertility)
7. Individuals with hypersensitivity to ingredients used in the investigational product(s)
8. Patients with serious infection (e.g., Sepsis) or active infection including localized infection
9. Patients with active tuberculosis
10. Patients with severe hepatopathy
11. Patients with an absolute neutrophil count (ANC) less than 500 cells/mm3
12. Patients with an absolute lymphocyte count (ALC) less than 500 cells/mm3
13. Patients who have hemoglobin levels less than 8 g/dL
14. Women who are pregnant or may be pregnant or lactating
15. Patients with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
16. Patients with nephropathy (BUN<8 or BUN>20 or Creatinine>1.5)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
AUCt of Chong Kun Dang Tofacitinib Tablet and XELJANZ 5Mg Tablet | Pre-dose (0 hour), post-dose 0.083, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
  Area under the Chong Kun Dang Tofacitinib Tablet / XELJANZ 5Mg Tablet concentration in blood-time curve from zero to final
Cmax of Chong Kun Dang Tofacitinib Tablet and XELJANZ 5Mg Tablet | Pre-dose (0 hour), post-dose 0.083, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours
  The maximum Chong Kun Dang Tofacitinib Tablet / XELJANZ 5Mg Tablet concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Bestian Hospital, Osŏng, South Korea

IPD SHARING:
Plan to Share IPD: No